CLINICAL TRIAL: NCT01919346
Title: Eculizumab for Prevention of Delayed Graft Function in Deceased Donor Kidney Transplantation
Brief Title: Eculizumab for Prevention of Delayed Graft Function (DGF) in Kidney Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on results from Alexion PROTECT DGF study
Sponsor: Heeger, Peter, M.D. (Individual)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-0920
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Delayed Graft Function; Kidney Transplantation; Complement Activity
Keywords: Kidney Transplantation; Delayed Graft Function
MeSH Terms: conditions — Delayed Graft Function | interventions — eculizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eculizumab (Experimental): Eculizumab 1200 mg (diluted in Sodium Chloride (NaCl) to 5mg/mL, volume = 240 mL) will be given intraoperatively at the time of transplantation prior to reperfusion of the renal allograft and again at 900 mg (diluted in NaCl to 5mg/mL, volume = 180 mL) 12-24 hours post-transplantation
  Interventions: Drug: Eculizumab
- Normal Saline (Placebo Comparator): Administered at same volume and time as Experimental arm
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Eculizumab
  Other Names: Soliris
  Arms: Eculizumab
Drug: Normal Saline
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to evaluate the efficacy of Eculizumab in the prevention of Delayed Graft Function following deceased donor kidney transplantation. Based on experimental data and supportive observations in humans associating complement gene upregulation with ischemic reperfusion (IR) injury, it is hypothesized that C5 cleavage is a key step in the pathogenesis of ischemic reperfusion injury following transplantation. It is further hypothesized that Eculizumab, a humanized monoclonal antibody that blocks C5 cleavage in humans will be an effective prophylactic agent to prevent IR injury in high risk recipients. This trial is a prospective, randomized study to test the efficacy of eculizumab vs. placebo given once at the time of transplantation and once again 24 hours later in preventing delayed graft function in first adult recipients of deceased donor kidneys.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Weight > 40 kg
* Male or Female
* Recipient of first deceased donor kidney
* Able to provide written informed consent
* Transplant candidate as per site specific guidelines
* Dialysis dependent renal failure (initiated more than 2 months prior to transplant)
* Recipients of kidneys defined as:

  1. Extended Criteria Donor (ECD) kidney with brain death: Kidney donors 60 years of age or older; or donors aged 50-59 years and have two of the following features: Hypertension, terminal serum creatinine > 1.5 mg/dL, or death from cerebrovascular accident (CVA), OR
  2. Standard Criteria Donor (SCD) kidney with actual cold ischemia time (CIT) 18 - 40 hours

Exclusion Criteria:

* Patient is planned to receive a multi-organ transplant
* Kidney from donor < 6 years of age
* Dual kidney transplant (from same donor, including en bloc)
* Living donor kidney transplant
* Recipients with donor-specific anti-HLA antibodies of more than 3,000 MFI
* Participation in another investigational drug study
* Recipient BMI > 40
* ABO incompatible
* DCD (donor with cardiac death) Donor
* Women who are pregnant or breast-feeding
* Women of child bearing potential who are unable or unwilling to use a medically acceptable form of contraception (defined as the use of oral, injected or implanted hormonal methods of contraception, intrauterine device (IUD)or intrauterine system (IUS), barrier methods of contraception (condom or occlusive cap with spermicidal foam/gel/film/cream/suppository)
* Patients with HBsAg-positive status, HCV infection, or HIV infection
* Patients with atypical hemolytic uremic syndrome (aHUS) or C3 glomerulonephritis (C3GN)
* Active bacterial or other infection which is clinically significant in the opinion of the investigator
* Patients with history of splenectomy
* Patients with history of meningococcal disease
* Patients allergic to or unable to tolerate Ciprofloxacin
* Patients unable or unwilling to receive vaccination against meningitis prior to study drug administration
* Patients with a known or suspected hereditary complement deficiency
* Patients with a history of cancer (other than non melanoma skin cancers) within the last five years
* Donors of more than 70 years of age
* Subjects with a psychiatric or physical illness which in the opinion of the Investigator would interfere with their ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Hemodialysis | 7 days post-transplantation
  The need of at least one dialysis treatment during the first 7 days after transplantation excluding: (i) requirement for a single dialysis session indicated for hyperkalemia (ii) hyperacute rejection, renal arterial and/or venous thrombosis, obstructive uropathy, recurrence of primary disease, and early thrombotic microangiopathy

SECONDARY OUTCOMES:
Estimated Glomerular Filtration Rate (GFR) | 6 months post-transplantation
  Estimated GFR as determined from the 4-variable MDRD (Modified Diet in Renal Disease) equation on days 7, 30, 90 and 180 post-transplantation
Hemodialysis | 8 weeks post-transplantation
  Number of dialysis sessions at 30 days and 8 weeks post-transplantation
Primary Non-function | 8 weeks post-transplantation
  The incidence of primary non-function (PNF) defined as the need for dialysis-dependency for more than 8 weeks
Graft Rejection | 6 months post-transplantation
  Incidence of graft rejection within 6 months
Patient Survival | 12 months post-transplantation
  Patient survival at 12 months post-transplantation
Graft Survival | 12 months post-transplantation
  Death censored graft survival at 12 months post-transplantation
Serum Creatinine | 3 days post-transplantation
  Change from baseline in serum creatinine and serum creatinine concentration at 24, 48 and 72 hours post-transplantation
Urine Output | 3 days post-transplantation
  Percentage of patients with total 24-hour urine output of more than 500 mL on post-transplantation days 2 and 3
Biomarkers | 6 months post-transplantation
  Absolute levels of biomarkers associated with acute renal injury
Qualified Delayed Graft Function (qDGF) | 7 days post-transplantation
  The incidence of qDGF defined as the requirement for dialysis for any reason in the first 7 days post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Heeger, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (5):
  - Yale - New Haven Hospital, New Haven, Connecticut
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania